CLINICAL TRIAL: NCT00293969
Title: A Randomized Clinical Trial Comparing Different Dosing Regimens of Intravenous Morphine in the Treatment of Adult Patients Presenting to the Emergency Department With Moderate to Severe Pain
Brief Title: A Trial Comparing Different Dosing Regimens of Morphine in Patients With Moderate to Severe Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-12-360
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2006-02-20 (Estimated); Status verified 2006-01

CONDITIONS: Pain
Keywords: Pain; Morphine
MeSH Terms: conditions — Pain | interventions — Morphine

INTERVENTIONS:
Drug: Morphine 0.1mg/kg versus morphine 0.15 mg/kg

SUMMARY:
RESEARCH QUESTION: In adult ED patients in whom the attending ED physician has decided to administer intravenous opiates, what is the difference in pain relief at 60 minutes in patients who are randomized to receive either weight-based IV morphine 0.1mg/kg or weight-based IV morphine 0.15 mg/kg?

HYPOTHESIS: In adult ED patients who receive IV morphine at a dose of 0.15/mg, more patients will report moderate to complete pain relief than patients receiving a dose of 0.1 mg/kg.

SIGNIFICANCE: If it is shown that morphine 0.15 mg/kg gives better pain relief to patients with comparable side effects when compared with morphine at a dose of 0.1 mg/kg, then we may be able to provide evidence to suggest that the higher dose should be used for adult ED patients under the age of 66 presenting with acute pain.

DETAILED DESCRIPTION:
RESEARCH QUESTION: In adult ED patients in whom the attending ED physician has decided to administer intravenous opiates, what is the between-group difference in before-after improvement in pain relief at 60 minutes in patients who are randomized to receive either weight-based IV morphine 0.1mg/kg or weight-based IV morphine 0.15 mg/kg?

HYPOTHESIS: In adult ED patients who receive IV morphine at a dose of 0.15/mg, more patients will report moderate to complete pain relief than patients receiving a dose of 0.1 mg/kg.

SIGNIFICANCE: If it is shown that morphine 0.15 mg/kg gives better pain relief to patients with comparable side effects when compared with morphine at a dose of 0.1 mg/kg, then we may be able to provide evidence to suggest that the higher dose should be used for adult ED patients under the age of 66 presenting with acute pain.

METHODS/DESIGN: Prospective, double blind, randomized clinical trial. Adult ED patients between the ages of 18 and 65 years of age in whom the attending ED physician has decided to administer parenteral opiates, will be randomized to receive either 0.1 mg/kg IV morphine (maximum dose of 10 mg) or 0.15mg/kg IV morphine (maximum dose of 15 mg). An on-line random plan generator (http://www.randomization.com) will be used to generate an allocation schedule. The allocation schedule will be fully documented with the reference citation of the pseudo-random number generator, the seed used to start the generation process, the number of treatments (2), the allocation ratio (1:1), the size and number of blocks, and a copy of the assignment list. The allocation schedule will be given to the Montefiore Department of Pharmacy where it will be used to determine the content of consecutively numbered vials with either the study doses of morphine. The Pharmacy Department will prepare and handle the vials in accordance with known stability data and labeled with expiration dates. They will provide the study with labeled packages containing the numbered vial, a label with the vial number to be attached to the patient's data collection instrument, an opaque envelope with the assignment group identified (to be used in the event of a clinical emergency that requires immediate determination of what the patient received) and a weight based dosing schedule for morphine. All patients will receive a bolus of morphine 0.1mg/kg at time 0. At 30 minutes, patients will receive the study drug which will contain either an additional 0.05mg/kg of morphine or placebo. After the initial morphine bolus and study drug, patients will have received either morphine 0.1 mg/kg (maximum of 10 mg) or 0.15 mg/kg (maximum of 15mg).

ELIGIBILITY:
Inclusion Criteria:

Patients 21 to 65 years of age presenting to the ED with pain of less than or equal to 7 days duration and deemed by the ED attending to require opioid analgesia are eligible for inclusion.

Exclusion Criteria:

Inability or unwillingness to provide informed consent, methadone use, use of other opioids or tramadol within 7 days, prior adverse reaction to morphine, chronic pain syndrome, alcohol intoxication, pregnancy or breast-feeding, systolic blood pressure <90 mm Hg, use of MAO inhibitors, and weight greater than 100 kg.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2005-03; Study Completion 2006-01

PRIMARY OUTCOMES:
The between-group difference in mean before-after difference in pain score at baseline and 60 minutes in patients randomized to receive either 0.10 mg/kg or 0.15 mg/kg morphine

SECONDARY OUTCOMES:
Between-group comparison of mean change in pain score from 30 min to 60 min
Comparison of between-group differences in pain relief scores
Patient satisfaction score
Adverse events at 30 and 60 minutes
Number of additional boluses of analgesics needed within 60 minutes for the two groups.
NRS pain score percent reduction at 60 min calculated as NRS pain score reduction from baseline to 60 min divided by baseline NRS score

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne J. Birnbaum, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center Emergency Department, The Bronx, New York, United States